CLINICAL TRIAL: NCT01736423
Title: A Long Term Study of YM060 in Female Patients With Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060-CL-703
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: YM060; Ramosetron; long term study; Diarrhea-predominant Irritable Bowel Syndrome; Female
MeSH Terms: interventions — ramosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Female Patients with D-IBS (Experimental)
  Interventions: Drug: YM060

INTERVENTIONS:
Drug: YM060 — oral
  Other Names: Ramosetron

SUMMARY:
To evaluate the efficacy and safety of YM060 once daily for female patients with diarrhea-predominant irritable bowel syndrome (D-IBS) for a long-term period (up to 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

Female patients who meet the following criteria:

1. Patients satisfying the Rome III Diagnostic Criteria
2. Patients whose ≥25% of stools were loose or watery and <25% of them were hard or lumpy stools
3. Patients who have abdominal pain or discomfort
4. Patients in whom after occurrence of IBS symptoms the following tests were conducted and in whom no organic changes were observed Pancolonoscopy or contrast enema

Exclusion Criteria:

Patients who meet any of the following criteria:

1. Patients with a history of surgical resection of the stomach,gallbladder, small intestine or large intestine
2. Patients with a history or current evidence of inflammatory bowel disease
3. Patients with a history or current evidence of colitis ischemic
4. Patients with concurrent infectious enteritis
5. Patients with concurrent hyperthyroidism or hypothyroidism
6. Patients with concurrent active peptic ulcer
7. Patients with other concurrent disease that may affect the digestive tract passage or large intestinal function or that is likely to interfere with proper assessment of IBS abdominal pain/discomfort

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Monthly responder rate of global assessment of relief of overall IBS symptoms | up to 52 weeks
Monthly responder rate of stool form normalization | up to 52 weeks
Monthly responder rate of global assessment of relief of abdominal pain/discomfort | up to 52 weeks
Monthly responder rate of global assessment of improvement of abnormal bowel habits | up to 52 weeks
Change in weekly average of scores of severity of abdominal pain/discomfort | up to 52 weeks
Change in weekly average of scores of stool form | up to 52 weeks
Change in weekly average of stool frequency | up to 52 weeks
Rate of days without urgency | up to 52 weeks
Rate of days without feeling of incomplete bowel movement | up to 52 weeks
Change in entire Japanese version of Irritable Bowel Syndrome Quality of Life (IBS-QOL-J) scores and pairwise IBS-QOL-J scores on the sub-scales | 4, 8, 12, 28 and 52 weeks

SECONDARY OUTCOMES:
Safety assessed through AEs and clinical laboratory values | up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu

REFERENCES:
- [Derived] Fukudo S, Kinoshita Y, Okumura T, Ida M, Hayashi K, Akiho H, Nakashima Y, Haruma K. Effect of ramosetron in female patients with irritable bowel syndrome with diarrhea: a phase III long-term study. J Gastroenterol. 2016 Sep;51(9):874-82. doi: 10.1007/s00535-016-1165-5. Epub 2016 Jan 22. PMID 26800997
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=060-CL-703